CLINICAL TRIAL: NCT06753838
Title: Choice of Anticoagulant for Primary Hemostasis Studies With PFA200® (Platelet Function Analyser)
Acronym: BAPAPFA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DE MAISTRE 2024
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hemostasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients requiring a PFA test for the diagnosis of Willebrand disease
  Interventions: Biological: Sampling of 3 additional BAPA tubes

INTERVENTIONS:
Biological: Sampling of 3 additional BAPA tubes — the 3 additional tubes will be taken at the same time as the blood sample taken for the routine PFA test

SUMMARY:
The PFA (platelet function analysis) test is prescribed for the exploration of primary hemostasis and the study of platelet-willebrand factor interaction. It is performed using citrated blood, with technical difficulties and frequent alarms that may be linked to the choice of anticoagulant (citrate). It is proposed to compare the results obtained with a conventional citrate tube and a BAPA tube, which is an anticoagulant used in clinical research and which blocks coagulation by another mechanism that would have less impact on blood platelets.

ELIGIBILITY:
Inclusion Criteria:

* Person having given their non-opposition
* Person of legal age
* Person receiving a haemostasis consultation at the haemophilia and haemorrhagic diseases treatment center followed by a blood sample with a PFA test prescribed by the doctor (the test is not added for the study).

Exclusion Criteria:

* persons under legal protection (curatorship, guardianship)
* persons subject to a court protection order
* pregnant, parturient or breast-feeding women
* adult incapable or unable to give consent
* minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a PFA test
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occlusion time measurement | at baseline
  Measurement of the occlusion times of the 2 cartridges (collagen/ADP and collagen/epinephrine) with the classic 0.109M citrate tube and the BAPA tube, with any PLC alarms and observation of the stained blood smears.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France